CLINICAL TRIAL: NCT02712866
Title: EARLY BIOMARKERS IN CIRCULATING α 4β7+ T CELLS TO PREDICT RESPONSE TO VEDOLIZUMAB IN INFLAMMATORY BOWEL DISEASE PATIENTS
Brief Title: Early Biomarkers in Circulating α 4β7 + T Cells to Predict Response to Vedolizumab in Inflamatory Bowel Disease Patients.
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Lucia Marquez, MD, PhD, Parc de Salut Mar
Other Study IDs: FIM-VED-2016-01
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with vedolizumab
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Administration of intravenous Vedolizumab in inflammatory bowel disease patients

SUMMARY:
Background: Infiltration of GI by T lymphocytes is a pathogenic mechanism both in ulcerative colitis (UC) and in Crohn's disease (CD). Vedolizumab (VDZ) is a humanized monoclonal antibody binding with high affinity to α4β7 integrin blocking α4β7+-MAdCAM-1 interaction, hence blocking a key step in GI lymphocytes T infiltration. VDZ has demonstrated a therapeutic effect in UC and CD. Investigators still lack of adequate biomarkers to predict clinical response to biological treatments, specially avoiding invasive procedures.

Objective: Study whether circulating CD4+ and CD8+ α4β7+ memory T lymphocytes and some of their surface markers might be molecular markers of response to VDZ treatment in patients with UC and CD.

Methods: Prospective (pilot) study including 24 adult IBD patients (12 UC patients and 12 CD patients (patients with fistulizing perianal disease will be excluded) with active disease and prior failure to anti-TNFα treatments starting treatment with VDZ. They will received VDZ in standard induction (300mg intravenously, 0-2-6 weeks) and maintenance schemes (300mg intravenously, every 8 weeks).

Epidemiological and clinical data from every patient will be recorded prospectively. Disease activity at weeks 0, 2, 6 and 14 weeks will be evaluated through validated clinical scores, biological parameters and fecal biomarkers.

At week 14 response to the treatment will be evaluated by ileocolonoscopy or enteroMRI.

Peripheral blood will be obtained from every patient at baseline, before the third infusion of VDZ (6th week) and before the first maintenance dose (14th week).

Blood lymphocytes will be isolated and multicolor flow cytometry will be performed on stored circulating memory T cells.

Percentage and absolute values of circulating CD4+ and CD8+ α4β7+ memory T lymphocytes as well as several surface markers related to their activation state (HLA-DR, CD25), Th17 phenotype (IL23R, CCR6, intracellular IL17A) and Th1 phenotype (INFγ)will be assessed on α4β7+ memory T cells.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis or Crohn's disease diagnosis established by Lennard-Jones criteria
* Clinically active disease confirmed by endoscopic or radiologic criteria Magnetic Resonance Image (MRI)
* >18 years of age
* Intolerant, refractory or secondary loss of response to anti-Anti-tumour necrosis factor (TNF) alfa treatment.

Exclusion Criteria:

* Crohn's disease with perianal disease
* Active Tuberculosis
* Current infections (including Clostridium difficile and Cytomegalovirus)
* History of cancer, including hematologic malignancy and solid tumours within 5 years before
* History of demyelinating disease
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24 adults with inflammatory bowel disease (12 Ulcerative colitis patients and 12 Chron Disease patients with active disease and prior failure to anti-TNFα treatments (inadequate response, loss of response, intolerance), starting treatment with Vedolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Surface and Th17 phenotype markers in T lymphocytes as response predictors | From drug administration until 14 weeks.

SECONDARY OUTCOMES:
Surface and Th17 phenotype markers in T lymphocytes as sustained remission predictors | From drug administration (week 14th) until 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No